CLINICAL TRIAL: NCT01478360
Title: A Randomized, Double-blind, Placebo Controlled, Multiple Dose Study to Evaluate the Safety, Tolerability, and Efficacy of Intravenous Administration of Secukinumab (AIN457) in Patients With Asthma Not Adequately Controlled With Inhaled Corticosteroids and Long Acting Beta-agonists.
Brief Title: Safety, Tolerability, and Efficacy of AIN457 in Patients With Uncontrolled Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Further investigations would require changes in study design; the use of different endpoints, a different IL-17 antibody or a different patient population.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457D2204
Record Dates: First submitted 2011-11-17; First posted 2011-11-23 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Asthma
Keywords: Asthma; Secukinumab; Therapeutic Uses; Respiratory; Lung; Pulmonary; inhaled; corticosteroids
MeSH Terms: conditions — Asthma; Respiratory Aspiration | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- AIN457 (Experimental): AIN457 10 mg/kg
  Interventions: Drug: AIN457 (secukinumab)
- Placebo (Placebo Comparator): Placebo intravenous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AIN457 (secukinumab) — Secukinumab intravenous injection
  Arms: AIN457
Drug: Placebo — Placebo intravenous injection
  Arms: Placebo

SUMMARY:
This study is a preliminary proof of efficacy study of AIN457 in patients with bronchial asthma that is poorly controlled with the current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with asthma >1 year duration diagnosed according to the GINA guidelines (GINA 2010).
* Daily treatment with > 1000μg beclomethasone dipropionate or equivalent, plus a long acting beta agonist for ≥ 3 months prior to Day 1, that has been stable for at least 4 weeks prior to screening.
* Asthma which is not adequately controlled on current treatment
* Peripheral blood eosinophil count < 400/μl at screening

Exclusion Criteria:

* Women of child-bearing potential unwilling to use effective contraception during the study and for 16 weeks after stopping treatment.
* Use of other investigational drugs at the time of screening, or within 30 days of screening.
* Smokers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Germany (5):
  - Novartis Investigative Site, Mainz, Germany
  - Novartis Investigative Site, Wiesbaden, Germany
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Großhansdorf
- United Kingdom (4):
  - Novartis Investigative Site, London, United Kingdom
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AIN457 | Placebo
Started | 31 | 15
PD (Pharmacodynamic) Analysis Set | 31 | 15
PK (Pharmacokinetics) Analysis Set | 31 (Serum samples were collected during the study and analyzed only for the AIN457 group) | 0
Completed | 29 | 12
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Administrative problems | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 | Placebo | Total
Number analyzed (Participants) | 31 | 15 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.8 (11.62) | 46.2 (10.40) | 48.6 (11.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 7 | 23
  Male | 15 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Improvement in the Severity of Asthma as Measured by Change in the Asthma Control Questionnaire (ACQ) Score
Description: The ACQ scores range from 0 to 6 with lower scores reflecting better asthma control. Without loss of generality, as Day 85 minus baseline (Visit 3) so that improvements in asthma control translate to negative change scores.
Time Frame: Baseline and 85 Days
Population: The Pharmacodynamics (PD) analysis set was used, and subjects were analyzed according to the treatment actually. The number of patients who had evaluable PD data at the particular PD assessment time point received.
Measure: Least Squares Mean (90% Confidence Interval); unit: Score
Arm/Group | AIN457 | Placebo
Number analyzed (Participants) | 29 | 13
Score | -0.173 [-0.425 to 0.079] | -0.007 [-0.380 to 0.365]
Statistical Analysis 1: Comparison: AIN457 vs Placebo; Test type: Superiority or Other; p = 0.5392, Mixed Models Analysis; Mean Difference (Net) = -0.166, 90% CI 2-sided [-0.617 to 0.285]

ADVERSE EVENTS:
Groups:
- AIN457 10 mg/kg: AIN457 10 mg/kg
- Placebo: Placebo
Arm/Group | AIN457 10 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/31 | 2/15
Other Adverse Events (participants affected / at risk) | 21/31 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 10 mg/kg (N=31) | Placebo (N=15)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 10 mg/kg (N=31) | Placebo (N=15)
TINNITUS (Ear and labyrinth disorders) | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1
ABDOMINAL RIGIDITY (Gastrointestinal disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 2
NAUSEA (Gastrointestinal disorders) | 2 | 4
VOMITING (Gastrointestinal disorders) | 1 | 3
CHILLS (General disorders) | 1 | 1
FATIGUE (General disorders) | 1 | 1
FEELING COLD (General disorders) | 0 | 1
VESSEL PUNCTURE SITE BRUISE (General disorders) | 0 | 1
CYSTITIS (Infections and infestations) | 2 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 2
NASOPHARYNGITIS (Infections and infestations) | 11 | 6
OTITIS EXTERNA (Infections and infestations) | 0 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
VIRAL INFECTION (Infections and infestations) | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 1 | 1
NAIL INJURY (Injury, poisoning and procedural complications) | 0 | 1
PERIORBITAL CONTUSION (Injury, poisoning and procedural complications) | 0 | 1
BODY TEMPERATURE INCREASED (Investigations) | 0 | 1
WEIGHT INCREASED (Investigations) | 0 | 1
IRON DEFICIENCY (Metabolism and nutrition disorders) | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1
DIZZINESS (Nervous system disorders) | 1 | 1
HEADACHE (Nervous system disorders) | 3 | 4
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 7 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 2
RASH (Skin and subcutaneous tissue disorders) | 0 | 1
XANTHOMA (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety